CLINICAL TRIAL: NCT03261830
Title: Antibiotics Usage in Pediatric Orthopaedic Percutaneous Surgery (APOPS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumit Gupta (Other)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Sponsor-Investigator, Sumit Gupta, Professor, Assistant Clinical - Department of Orthopaedic Surgery, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2008610
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Supracondylar Humerus Fracture; Post Operative Wound Infection
Keywords: Antibiotic; Pediatric
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Clindamycin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in that one group receives one dose of pre-operative antibiotics or one that does not.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization envelops will be created. Attending surgeons/Investigators will be blinded. Participant will be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pre-operative Antibiotics (Active Comparator): Patients randomized to preoperative antibiotics will receive 25mg/kg cefazolin IV up to 1g or clindamycin 10mg/kg up to 600mg IV in cases of documented allergy to cefazolin.
  Interventions: Drug: Cefazolin; Drug: Clindamycin
- Saline Placebo (Placebo Comparator): Patients randomized to the no-antibiotic group will receive a saline placebo. This placebo will consist of a 10 mL pre-filled syringe of normal saline.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Cefazolin — Primary intervention
  Arms: Pre-operative Antibiotics
Drug: Clindamycin — For use in Pre-operative Antibiotics arm in cases of documented allergy to primary intervention.
  Arms: Pre-operative Antibiotics
Drug: Saline — Placebo Intervention
  Arms: Saline Placebo

SUMMARY:
The aim of this study is to determine if antibiotics affect the outcome after percutaneous surgery for pediatric supracondylar humerus fractures. The patient population will be recruited from the cohort presenting to Women and Children's Hospital for percutaneous fixation of pediatric supracondylar humerus fractures who meet the eligibility criteria and consent to taking part in the study. Patients will be followed up for 3-6 weeks depending on age, and will be evaluated on the presence or absence superficial or deep infection, Visual Analog Scale pain scores, time to healing, need for repeat casting, and loss of fixation.

DETAILED DESCRIPTION:
This patient population will be recruited from the cohort presenting to Women and Children's Hospital for percutaneous fixation of pediatric supracondylar humerus fractures. Participants will be asked to assent to take part in the study and their parents or guardian will be asked to sign an informed consent. Patients will be randomized to a treatment group that receives one dose of pre-operative antibiotics or one that does not. Patients randomized to preoperative antibiotics will receive 25mg/kg cefazolin IV up to 1g or clindamycin 10mg/kg up to 600mg IV in cases of documented allergy to cefazolin. Patients randomized to the no-antibiotic group will receive a saline placebo. The resident, anesthesiologist, circulating nurse and other operating room staff will be instructed to not reveal the patient's randomization to the attending physician so as not to interfere with blinding.

The patient will then undergo closed reduction percutaneous pinning of supracondylar humerus fracture. Final AP and lateral fluoroscopic images in the case will be taken. The patient will be discharged from the hospital when pain is controlled with standard oral pain medications and all goals of inpatient management have been achieved. No patients will receive post-operative antibiotics regardless of randomization group as is the existing standard of care. Patients will be scheduled to follow up in 3-6 weeks depending on age. At that time the cast will be removed and AP and lateral radiographs will be used to assess healing. The pins will be removed in clinic and a soft dressing applied to the elbow region.

In cases of excessive pain or cast loosening the patient may be seen in clinic earlier with radiographs and physical exam as indicated. If the attending physician determines that a deep or superficial infection is present at any time during the treatment period the patient will be categorized as infected. If no infection is detected at an earlier-scheduled appointment the patient will be recasted and instructed to follow up as previously scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Age<14 years
* Open growth plates
* Gartland type II or III extension type fracture of the distal humerus OR Flexion type fracture of the distal humerus

Exclusion Criteria:

* Need for open reduction
* Need for antibiotics due to other injuries or conditions during the entire study period
* Immunosuppression
* History of malignancy or metabolic bone disease
* Open fractures
* Pre-existing Infection
* Intra-operative breech of sterile technique

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Gupta, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States

REFERENCES:
- [Derived] Gupta SK, Esposito ER, Phillips R, Schwab PE, Leary EV, Hoernschemeyer DG. Effect of Antibiotic Prophylaxis on Infection Rates in Pediatric Supracondylar Humerus Fractures Treated with Closed Reduction and Percutaneous Pinning: A Prospective Double-Blinded Randomized Controlled Trial. J Am Acad Orthop Surg. 2024 May 1;32(9):410-416. doi: 10.5435/JAAOS-D-23-00795. Epub 2024 Feb 28. PMID 38422496

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-operative Antibiotics | Saline Placebo
Started | 82 | 78
Completed | 82 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-operative Antibiotics | Saline Placebo | Total
Number analyzed (Participants) | 82 | 78 | 160
Age, Continuous [Mean (Full Range); unit: Years] | 5.9 [1.1 to 11.7] | 5.5 [1.3 to 12.5] | 5.67 [1.1 to 12.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 47 | 87
  Male | 42 | 31 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Presence of Post-Operative Infection
Description: The primary outcome measure will be the presence of infection as judged by the blinded attending surgeon at the time of cast removal. A superficial infection is defined as a clinical diagnosis based on increased erythema, granulation tissue or purulence at the pin sites that resolves with a short course of oral antibiotics. A deep infection is defined as the presence of septic arthritis or osteomyelitis requiring return to the operating room for debridement or a prolonged course of IV antibiotics. If the attending physician determines that a deep or superficial infection is present at any time during the treatment period the patient will be categorized as infected.
Time Frame: Six weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Antibiotics | Saline Placebo
Number analyzed (Participants) | 82 | 78
Participants | 2 | 2

2. Secondary Outcome: Visual Analog Pain Scale
Description: Presented as a 100mm horizontal line on which the patient's pain intensity is represented by a point between two extremes of "no pain at all" = 0 and "worst pain imaginable" = 100.
Time Frame: Three to Six Week Follow Up
Population: The VAS data was not collected and will therefore not be reported.
Arm/Group | Pre-operative Antibiotics | Saline Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Fractures Fully Healed
Description: Time to healing/fractures fully healed was measured by the review of AP and Lateral radiographs at the first follow-up and considered healed if at least 3 cortices had callus. This outcome measure is reported as the number of participants in each group with fully healed fractures at the designated time point.
Time Frame: Three to Six Week Follow Up
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Antibiotics | Saline Placebo
Number analyzed (Participants) | 82 | 78
Participants | 82 | 78

4. Secondary Outcome: Number of Participants With a Need for Repeat Casting
Description: The need for repeat casting can be due to excessive pain or loosening of the cast.
Time Frame: Three to Six Weeks Follow Up
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Antibiotics | Saline Placebo
Number analyzed (Participants) | 82 | 78
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Experiencing Loss of Fixation
Description: Loss of fixation (stabilization) refers to a situation where the fixation of the fracture become compromised.
Time Frame: Three to Six Weeks Follow Up
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Antibiotics | Saline Placebo
Number analyzed (Participants) | 82 | 78
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 6 weeks or until the fracture is healed.
Description: There is no difference in the definition of adverse event and/or serious adverse event from that of clinicaltrials.gov.
Arm/Group | Pre-operative Antibiotics | Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/78
Serious Adverse Events (participants affected / at risk) | 1/82 | 0/78
Other Adverse Events (participants affected / at risk) | 0/82 | 1/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-operative Antibiotics (N=82) | Saline Placebo (N=78)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-operative Antibiotics (N=82) | Saline Placebo (N=78)
Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Superficial infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03261830/Prot_000.pdf